CLINICAL TRIAL: NCT05271838
Title: Nutritional Therapy for Patients With Acute Severe Ulcerative Colitis (ASUC) Treated With High-dose Steroids - a Special Focus on Protein and Magnesium.
Brief Title: Protein and Magnesium in Ulcerative Colitis
Acronym: PAMUC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Christian Hvas, Associate professor, MD PhD, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-363-21
Record Dates: First submitted 2022-02-17; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Inflammatory Bowel Diseases; Colitis, Ulcerative; Magnesium Deficiency; Nutritional Deficiency; Protein Deficiency
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Magnesium Deficiency; Malnutrition; Protein Deficiency | interventions — Diet, High-Protein

STUDY DESIGN:
Intervention Model Description: At baseline patients are randomized to either a dietary protein intake of 2 g/kg/day (achieved by nutritional counseling and protein supplementations) or standard care (No nutritional counseling or protein recommendation are given) under admission and three weeks after discharge.
  Furthermore patients with a magnesium retention level >25% are further randomized to receive either magnesium acetate oral mixture (0,5 mmol/ml) 20 ml x 3 daily (30 mmol/day) or not receiving magnesium supplement for three weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High protein diet (Experimental): High protein diet (2/g/kg/day)
  Interventions: Dietary Supplement: High-protein diet (2 g/kg/day)
- Standard Nutritional care (No Intervention): Standard nutritional care.
- Magnesium (Experimental): Magnesium oral supplementation
  Interventions: Dietary Supplement: Magnesium acetate mixture (30 mmol/ml)
- Standard: No magnesium supplementation (No Intervention): No supplementation

INTERVENTIONS:
Dietary Supplement: Magnesium acetate mixture (30 mmol/ml) — Patients with a magnesium retention test >25% and randomized to intervention receive magnesium acetate oral mixture (30 mmol/ml) 20 ml x 3/day for a period of three weeks.
  Arms: Magnesium
Dietary Supplement: High-protein diet (2 g/kg/day) — Nutritional counseling and protein supplementation to establish an intake of 2 g protein kg/day during admission and three weeks after discharge.
  Arms: High protein diet

SUMMARY:
The aim of the study is to improve the quality of nutritional therapy for patients admitted with Acute Severe Ulcerative Colitis (ASUC) treated with high-dose steroids. This study consists of two randomized interventions and one observational part regarding protein, magnesium, and metabolic stress. First an interventional part aims to explore the effect of a high-protein diet during and after admission on different parameters regarding protein turnover.Second the study aims to explore the degree of magnesium depletion in ASUC. In case of magnesium depletion, the study aims to investigate whether oral magnesium supplementation can regain body stores of magnesium. Last the study aims to observe the degree of metabolic stress, including, the degree of insulin resistance, in ASUC during admission and under treatment with high-dose steroids compared to three weeks after discharge.

DETAILED DESCRIPTION:
Patients with Acute Severe Ulcerative Colitis (ASUC) may have an altered protein turnover due to inflammation, reduced dietary intake and/or accelerated protein loss. Despite this the level of dietary protein needed to maintain nitrogen balance has never been described in patients with ASUC. Clinical symptoms of ASUC include frequent and bloody diarrhea which alone or simultaneous with a risk of reduced dietary intake and weightloss can lead to magnesium depletion. Magnesium depletion can cause severe symptoms including cardiac arrhythmia and neuromuscular dysfunction which might worsen the disease further. The prevalence of magnesium depletion in ASUC has never been described and furthermore it is not known whether oral supplementation are able to reverse the condition in patients with ASUC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Cognizant
* Must speak or read Danish or participate in relevant communication in interpreting or translating the study material.
* Diagnosed with Acute Severe Ulcerative Colitis (ASUC) (documented in the patient journal)
* Admitted at "Lever-, Mave-, og Tarmsygdomme/ LMT" at Aarhus University Hospital and in medical treatment with high-dose intravenous steroid (Solumedrol 40 mg x 2 daily)

Exclusion Criteria:

* Pregnant and/or lactating women
* Plasma creatinine > 200 µmol/L (protein intervention only)
* Patients receiving tube- or parenteral feeding (protein intervention only)
* Receiving any kind of magnesium supplementation 6 months prior to inclusion (magnesium intervention only)
* Diagnosed with Type 1 or Type 2 Diabetes Mellitus (observational part only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
24 hour urine carbamide (mmol/d) | 5 days
  Change in 24 hour urine carbamide (mmol/d) from baseline (day 0) to first follow-up (day 5)

SECONDARY OUTCOMES:
24 hour urine carbamide (mmol/d) | 4 weeks
  Change in 24 hour urine carbamide (mmol/d) between baseline (day 0) and at week 4
24 hour urine creatinine (mmol/d) | 0, follow up 1 (day 5) and week 4
  Change in 24 hour urine creatinine (mmol/d)
24 hour urine magnesium (mmol/d) | 3 weeks
  Change in 24 hour urine magnesium (mmol/d) between follow up 1 (day 5) and after three weeks.
Magnesium retention % | 3 weeks
  Change in magnesium retention (%) between follow up 1 (day 5) until after three weeks.
Quality of life (QOL) questionaire (SIBDQ) | 3 weeks
  Change in QOL-score patient administered QOL-scoring system - The short bowel inflammatory bowel disease questionaire (SIBDQ) between follow-up 1 (day 5) and after three weeks.
Quality of life (QOL) questionaire (Hjortswang index) | 3 weeks
  Change in QOL-score patient administered QOL-scoring system - Hjortswang index between follow-up 1 (day 5) and after three weeks.
Fat free mass (FFM) (kg) | 4 weeks
  Change in FFM (kg) between baseline and after four weeks. Measured after minimum 6 hours of fasting by Bioimpedance spectroscopy.
Resting Energy Expenditure (REE) | 4 weeks
  Change in REE between baseline and after four weeks. Measured after minimum 6 hours of fasting by indirect calorimetry.
Body weight (kg) | 4 weeks
  Change in body between baseline and after four weeks. Measured after minimum 6 hours of fasting by Bioimpedance spectroscopy.
plasma carbamide (mmol/l) | 0, follow-up 1 (day 5) and week 4
  Change in plasma carbamide (mmol/l) measured at baseline, follow up 1(day 5) and at week 4.
plasma magnesium (mmol/l) | 4 weeks
  Change in plasma magnesium (mmol/l) between follow-up 1 (day 5) and at week 4
plasma albumin (g/L) | 4 weeks
  Change in plasma albumin (mmol/l) between follow-up 1 (day 5) and at week 4
plasma insulin (pmol/l) | 4 weeks
  Change in plasma insulin (pmol/l) between baseline and week 4
plasma c-peptide (pmol/l) | 4 weeks
  Change in plasma c-peptide (pmol/l) between baseline and week 4
Fasting blood glucose (mmol/l) | 4 weeks
  Change in fasting blood glucose (mmol/l) after a minimum of 6 hours fasting between baseline and week 4
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)-score | 4 weeks
  Change in HOMA-IR-score between baseline and week 4
Creatinine-clearance (mL/min) | 0, follow-up 1 (day 5) and week 4
  Change in creatinine-clearance (ml/min)

OTHER OUTCOMES:
Protein intake (g/kg/day) | Week 1 and week 4
  Assessment of dietary protein intake during admission and after discharge by patient dietary registration schedules and supplemented by 24-h recall during admission.
Energy intake (kcal/day) | Week 1 and week 4
  Assessment of dietary intake during admission and after discharge by patient dietary registration schedules and supplemented by 24-h recall during admission.
Physical activity level (hours/week) | 4 weeks
  Patients are asked about habitual physical activity level (hours/week) in the period before admission and physical activity level within 3 weeks after discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided